CLINICAL TRIAL: NCT06738745
Title: A Phase II Study of HRS-2189 Combined HRS-5041 in Metastatic Prostate Cancer
Brief Title: Study of HRS-2189 Combined HRS-5041 in Prostate Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ding-Wei Ye, Chief physician, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRPC-MUL-IIT-HRS2189-HRS5041
Record Dates: First submitted 2024-11-22; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer Metastatic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HRS-2189 + HRS-5041 (Experimental): All subjects enrolled will receive HRS-2189 + HRS-5041 combination therapy.
  Interventions: Drug: HRS-2189; Drug: HRS-5041

INTERVENTIONS:
Drug: HRS-2189 — HRS-2189
Drug: HRS-5041 — HRS-5041

SUMMARY:
Our study is aimed to evaluate the efficacy and safety of HRS-2189 combined with HRS-5041 in metastatic prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18 years to 80 years old (including boundary values), male subjects;
* ECOG PS Score: 0~1;
* Histologically or cytologically confirmed prostate adenocarcinoma, and no prior diagnosed as neuroendocrine carcinoma or small cell carcinoma;
* Disease progression when enrolled in the study;
* Confirmed metastatic disease by CT/MRI/99mTc radioactive bone scan;
* Subjects must have a life expectancy ≥ 3 months;
* Adequate organ function and marrow function (no corrective treatment within 14 days before first dose);
* Male subjects who have partner of childbearing potential should agree to take action of contraception and avoid to donate sperm;
* Willing and able to provide written informed consent and comply with the requirements and restrictions in the protocol.

Exclusion Criteria:

* Known existence of CNS metastasis or meningeal metastasis, or known history of primary CNS tumor;
* Severe bone injury caused by bone metastasis identified by investigators, including uncontrolled severe bone pain, pathological bone fracture at the important part and spinal cord compression having occurred for the last 6 months or expected to occur in the near future;
* Existence of third space fluid that is not well controlled by effective methods, e.g. drainage;
* Has received antitumor surgery, radiotherapy, chemotherapy, targeted therapy, immunological therapy or attenuated live vaccine within 4 weeks before first dose of study therapy (6-week washout period for bicalutamide);
* Has been enrolled in other clinical trials within 4 weeks before first dose of study therapy;
* Use of other antitumor treatment during the study;
* Damage caused by any prior anti-tumor treatment has not recovered to ≤ grade 1 or criteria specified by this study (per NCI-CTCAE 5.0; except alopecia or other tolerable adverse events identified by investigators);
* Uncontrolled hypertension, or prior hypertensive crisis or history of hypertension;
* Existence of arterial/venous thrombotic event within 6 months before first dose, such as cerebrovascular accidents (including transient ischemic attack, cerebral haemorrhage and cerebral infarction), deep venous thrombosis and pulmonary embolism;
* Existence of one of multiple factors that affect oral medication (such as inability to swallow, chronic diarrhea and bowel obstruction), or active gastrointestinal disease or other diseases which may obviously affect distribution of drug absorption, metabolism or excretion;
* Has active hepatitis B (HBsAg-positive and HBV DNA≥500 IU/mL), hepatitis C (positive for HCV antibody and HCV RNA above ULN) and hepatic cirrhosis;
* Has an active infection requiring antibiotics, antiviral or antifungal treatment, or pyrexia >38.5℃ of unknown origin during the screening period before first dose of study therapy (patients with pyrexia due to cancer could be enrolled determined by investigator);
* Subjects with innate or acquired immunodeficiency (such as HIV infection); Known history of allogeneic organ transplantation or hematopoietic stem cell transplantation;
* Other malignancy within prior 3 years before first dose of study therapy, except curatively treated cancer, including radical therapy-treated skin basal cell carcinoma or skin squamous cell carcinoma, papillary thyroid carcinoma, or any type of in situ carcinoma with complete excision, such as in situ cancer of the cervix, ductal carcinoma in situ of breast;
* Hypersensitivity to study therapy or any of its excipients;
* Uncontrolled cardiovascular clinical symptom or disease within 6 months before first dose of study therapy;
* Other conditions that might influence the study and analysis of results in the opinion of the investigator.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-12-31 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
PSA50 | up to 2 years
  PSA50 is the percentage of evaluable patients with ≥50% decline in PSA level, measured at baseline and the time point of every 4 weeks in efficacy analysis set.

SECONDARY OUTCOMES:
PSA30 | up to 2 years
  PSA30 is the percentage of evaluable patients with ≥30% decline in PSA level measured at baseline and the time point of every 4 weeks in efficacy analysis set.
Time to PSA progression | up to 2 years
  The definition is the time from the date of first dose until the date of first PSA progression or death (by any cause in the absence of progression). PSA progression is per PCWG3 criteria and newest version of CSCO guideline as follows: 1) if PSA level declines from baseline, PSA level is ≥25% increase from baseline and ≥1 ng/ml, which needs to be confirmed after at least 4 weeks; 2) if PSA level has not declined from baseline, PSA level is ≥25% increase from baseline and ≥1 ng/ml after at least 12 weeks from the date of first dose.
ORR by investigator | up to 2 years
  ORR is the percentage of evaluable patients with a confirmed investigator-assessed response of CR (complete response) or PR (partial response) per RECIST v1.1, and measured at baseline and the time point of every 8 weeks in first 16 weeks, at the time point of every 12 weeks after first 16 weeks.
DCR by investigator | up to 2 years
  DCR is the percentage of evaluable patients with a confirmed investigator-assessed response of CR (complete response), PR (partial response) or SD (stable disease) per RECIST v1.1, and measured at baseline and the time point of every 8 weeks in first 16 weeks, at the time point of every 12 weeks after first 16 weeks.
DoR | up to 2 years
  DoR is the time from the date of first detection of objective response (which is subsequently confirmed) until the date of objective radiographic disease progression.
rPFS | up to 2 years
  rPFS is the time from the date of first dose until the date of objective radiographic disease progression or death (by any cause in the absence of progression) per RECIST v1.1 and PCWG3 criteria.
Time to next skeletal-related event | up to 2 years
  The definition is the time from the date of first dose until the date of next skeletal-related event. Skeletal-related events include radiotherapy or surgery to the bone, pathological bone fracture, spinal cord compression, or changing anti-tumor treatment in order to relieve bone pain.
OS | up to 2 years
  OS is the time from the date of first dose until the date of death by any cause.
Percentage of participants who experience an adverse event [Safety and Tolerability] | From the time of informed consent provided to 30 days after the last dose of study therapy
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. Percentage of participants who experience an adverse event and discontinue study drug due to an AE.

CONTACTS AND LOCATIONS:
Overall Officials: Dingwei Ye, Chief physician, Principal Investigator — Fudan University
Locations (1):
- Fudan Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No